CLINICAL TRIAL: NCT00624260
Title: Impact of PET Scan on the Curative Strategy of Colo-rectal Cancers : A Randomized Study
Acronym: ITEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: P070142
Record Dates: First submitted 2008-02-15; First posted 2008-02-27 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Recurrence; Positron Emission Tomography; Colorectal Cancer with high risk of recurrence stage III; Colorectal Cancer with high risk of recurrence stage IV; T4N0M0 operated in emergency( because of perforation)
MeSH Terms: conditions — Colorectal Neoplasms; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 2 (Active Comparator): Usual follow up : Pet-TDM for current indication (high isolated markers or before a metastasis curative resection)
  Interventions: Other: PET-TDM for current indication
- 1 (Experimental): Semi-annual systematic PET-TDM (M6, M12, M18, M24, M30 and M36 after initial surgery)
  Interventions: Other: semi-annual systematic PET-TDM

INTERVENTIONS:
Other: semi-annual systematic PET-TDM — semi-annual systematic PET-TDM
  Arms: 1
Other: PET-TDM for current indication — PET-TDM for current indication (high isolated markers or before a metastasis curative resection)
  Arms: 2

SUMMARY:
The risk of recurrence in stage III and IV of colorectal cancers (CRC) is high during the three years following the tumoral resection with curative aim. Therefore, a prolonged follow-up and an intense monitoring are recommended to detect these recurrences precociously. Nevertheless, current consensual morphological and biological examinations are not very contributory, of difficult interpretation and expensive. The metabolic imagery in tomoscintigraphy by emission of positron coupled with the scanner, called PET-TDM, allows to identify more specifically recurrences, analyzes the whole body, detects hepatic metastasis more precociously and give some benefice for early diagnosis of lymph nodes recurrence. The principle purpose of this study is to evaluate if the systematic follow-up per PET-TDM allows detecting more often recurrences accessible to a curative surgery. We make the hypothesis that the systematic practice of PET- tomodensitometry (TDM) during the follow-up of CRC allows to decrease non curative recurrences appearance during the 3 years follow-up after a curative surgery.

DETAILED DESCRIPTION:
Patients will be randomized in two groups: one (PET-TDM group) including a semi-annual systematic PET-TDM during usual follow-up (M6, M12, M18, M24, M30 and M36 after initial surgery) and the second (control group) in which one PET-TDM will be realized only for current indication (high isolated markers or before a metastasis curative resection) during usual follow-up. Will be included patients with a high risk of recurrence of a colorectal tumor N+ or M+ completely removed (R0 or R1) or tumor stage 4, no regional lymph node metastasis, no distant metastasis (T4N0M0) operated in emergency (tumoral perforation).

Patients will be followed-up during 3 years since the date of initial surgery. Conventional follow-up will be performed by consensual recommendations for all the patients. In the case of detecting a recurrence, the adapted treatment (surgery or chemotherapy or both) with curative aim will be implemented and the follow-up will be carried out in its term or death. In the case of non curable recurrence, the follow-up will be carried out in its term or death, and the PET-TDM will not be realised any more.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a removed colorectal adenocarcinoma since less than 6 months, in total remission and for whom a monitoring is necessary to detect recurrences precociously.
* Patients with a removed colorectal tumour which is histologically proved and classified N+ and/or M+ (stage III or IV). Hepatic and/or pulmonary metastasis would have been totally removed since less 6 months before inclusion.
* Patients with a T4N0M0 tumour and operated in emergency (because of a tumoral perforation) can be included. (suppressed by amendment 1)
* 2 before criteria have been replaced by : Patients with colorectal adenocarcinoma which is histologically proved and classified stage II perforated, III or IV, totally removed, in total remission,
* if no metastatic, removed surgery must have been done since less 6 months;
* if metastatic, all metastasis would have been removed, the last surgery dating less 6 months.(amendment 1)
* Casual extension check-up would have been realized before initial surgery or during a period of 6 months after surgery performed in emergency.
* informed consent signed
* Age ≥ 18 years
* Patient in ability to undergone hepatic or pulmonary resection in case of recurrence during the follow-up (ECOG ≤ 2)
* Willingness to control visits

Exclusion Criteria:

* pregnant or breast feeding women, or with a reproductive potential and no practicing an effective method of contraception during the second part of ovarian cycle ( PET is realised during the first part of ovarian cycle)
* Cancer stage I or II (except T4 operated in emergency) or IV without possibility to remove metastasis or R2 after surgery.
* Performance status contraindicating a hepatic or pulmonary surgery in case of recurrence.
* Patients likely to undergone chemotherapy, surgery or radiotherapy during 2 weeks before PET-TDM.
* Other progressive tumoral affection known, or colorectal cancer in progression.

  • (Bad compliance to the study procedure.)(suppressed by amendment 1)
* Not balanced diabetes. (added by amendment 1)
* Patients included in others clinical trials of imagery.
* Inability to provide informed consent signed.
* No social assurance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2008-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with a non removable recurrence | at the end of the study

SECONDARY OUTCOMES:
Survival without non removable tumor | At the end of the study
Overall survival | At the end of the study
Cost of the strategy | At the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Iradj Sobhani, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- CHU Henri Mondor, Créteil, France

REFERENCES:
- [Derived] Sobhani I, Itti E, Luciani A, Baumgaertner I, Layese R, Andre T, Ducreux M, Gornet JM, Goujon G, Aparicio T, Taieb J, Bachet JB, Hemery F, Retbi A, Mons M, Flicoteaux R, Rhein B, Baron S, Cherrak I, Rufat P, Le Corvoisier P, de'Angelis N, Natella PA, Maoulida H, Tournigand C, Durand Zaleski I, Bastuji-Garin S. Colorectal cancer (CRC) monitoring by 6-monthly 18FDG-PET/CT: an open-label multicentre randomised trial. Ann Oncol. 2018 Apr 1;29(4):931-937. doi: 10.1093/annonc/mdy031. PMID 29365058